CLINICAL TRIAL: NCT05663281
Title: Thrombus Imaging and Treatment Analytics in Neurology
Acronym: Titan
Status: Recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Jinhao Lyu, Attending physician, Chinese PLA General Hospital
Other Study IDs: 301Titan
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Thrombus, Brain; Thrombosis
Keywords: Thrombus; Neuroimaging; High-resolution vessel wall imaging; Cerebral ischemia; Cerebral artery
MeSH Terms: conditions — Intracranial Thrombosis; Thrombosis; Brain Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: thrombus imaging appearance — Imaging appearance of intracranial and/or extracranial arterial thrombus

SUMMARY:
In the present study, the investigators use high-resolution MR vessel wall imaging, and select patients with cerebral and cervical artery occlusion to investigate the relationship between the imaging appearance of thrombus and the various outcome of recanalization treatment.

DETAILED DESCRIPTION:
Cerebral ischemic stroke resulting from thrombosis causes high disability and mortality. There are few biomarkers to evaluate arterial thrombophilia until now. Previous studies have demonstrated that atherosclerotic plaque rupture and erosion are major etiologies initiating thrombosis. Based on previous works targeting the role of plaque and blood flow in cerebrovascular disease, in the present study, the investigators use high-resolution MR vessel wall imaging, and select patients with cerebral and cervical artery occlusion to explore the relationship between the imaging appearance of thrombus and the various outcome of recanalization treatment. The study's objective was to solve the challenges in the mechanism of thrombus features and the outcome of recanalization therapy, thus helping improve the primary and secondary prevention of cerebrovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Extracranial and/or intracranial artery occlusion confirmed by angiography
* Available for magnetic resonance high-resolution vessel wall imaging
* Written informed consent obtained

Exclusion Criteria:

* Extracranial and/or intracranial artery mild to moderate stenosis
* Pregnant women
* Restenosis or occlusion after artery stenting placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who are confirmed to have extracranial and/or intracranial artery occlusion
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Successful Recanalization | 1-3 Years
  Antegrade blood flow through the recanalized portion was assessed by thrombolysis in myocardial infarction (TIMI) score or thrombolysis in cerebral infarction (TICI) score. TIMI≥2 or TICI≥2b was defined as successful recanalization.
Ischemic Stroke Occurrence | 1-3 Years
  Ischemic stroke occurrence during follow-up period which was confirmed by neuroimaging

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | 1-3 Years
  hemorrhagic or ischemic stroke after recanalization treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China